CLINICAL TRIAL: NCT06333249
Title: A Phase 1/2 Open-Label Dose Escalation Study to Evaluate the Safety and Efficacy of AGTC-501 (rAAV2tYF-GRK1-RPGR) and a Phase 2 Randomized, Controlled, Masked, Multi-center Study Comparing Two Doses of AGTC-501 in Male Subjects With X-linked Retinitis Pigmentosa Confirmed by a Pathogenic Variant in the RPGR Gene
Brief Title: A Study Comparing Two Doses of AGTC-501 in Male Subjects With X-linked Retinitis Pigmentosa Caused by RPGR Mutations (SKYLINE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGTC-RPGR-001 SKYLINE
Record Dates: First submitted 2024-02-16; First posted 2024-03-27 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP; retinal degeneration; RPGR; adeno-associated virus; gene therapy; AAV
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: The purpose of the Phase 2 study is to evaluate the efficacy, safety, and tolerability of two doses of AGTC-501 in male subjects between 8 - 50 years of age (inclusive) with XLRP genetically confirmed by at least one pathogenic variant in the RPGR gene.
  Approximately 12 subjects who meet the inclusion criteria, will be randomized in a 1:1 ratio to 1 of 2 treatment groups. Each subject will receive the assigned dose of AGTC-501 in the study eye; no treatment will be administered in the fellow eye. As treatment outcomes in pediatric vs. adult subjects may differ, randomization to dose groups will be stratified by age.
  Each subject will receive a central subretinal injection of AGTC-501 at the assigned dose in the central macula of the study eye.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Phase 2 study is a masked study; therefore, neither the investigator nor the subject will know the dose assignment. Both the subject and the investigator will know which eye received treatment.
  Masking will continue until the Month 12 data analysis is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Group (Experimental): Male subjects at least 8 y/o treated with a lower dose (Dose 2 in RPGR-001 Horizon Phase 1/2 study) of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR
- High Dose Group (Experimental): Male subjects at least 8 y/o treated with a higher dose (Dose 5 in RPGR-001 Horizon Phase 1/2 study) of rAAV2tYF-GRK1-RPGR study drug.
  Interventions: Biological: rAAV2tYF-GRK1-RPGR

INTERVENTIONS:
Biological: rAAV2tYF-GRK1-RPGR — Adeno-associated virus vector expressing a human RPGR gene

SUMMARY:
This study will evaluate the safety and efficacy of a recombinant adeno-associated virus vector (rAAV2tYF-GRK1-RPGR) in patients with X-linked retinitis pigmentosa caused by RPGR mutations.

DETAILED DESCRIPTION:
Approximately 12 participants, who were not part of the Phase 1/2 (HORIZON) study, will be enrolled into the dose expansion portion of the study. These participants will be randomized in a 1:1 ratio to 1 of 2 treatment groups (i.e., Group 1 [low dose] and Group 2 [high dose]). Each participant will receive the assigned dose of AGTC-501 in one eye on a single occasion.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent or assent (per local regulation), prior to the conduct of any study-related procedure. Subjects who provide assent must have a parent, guardian, or legal representative provide written informed consent.
* Be between 8 and 50 years of age (inclusive) at the time of informed consent and assent (as applicable).
* Be male and have at least one documented pathogenic or likely pathogenic variant in the RPGR gene
* Have a clinical diagnosis of XLRP.
* Have a BCVA no better than 75 letters and no worse than 35 letters based on an ETDRS chart at each screening visit.
* Be able to perform all tests of visual and retinal function and structure in both eyes based on the subject's reliability, and fixation, per the investigator's discretion.
* Have detectable baseline mean macular sensitivity measured by (MAIA) microperimetry, as determined by the investigator and confirmed by the Central Reading Center (CRC).
* Have detectable EZ line in both eyes as assessed by SD-OCT and confirmed by the CRC.

Exclusion Criteria:

* Have other known disease-causing mutations documented in the subject's medical history or identified through a retinal dystrophy gene panel, that in the opinion of the investigator would interfere with the potential therapeutic effect of the study agent or the quality of the assessments.
* For subjects with herpes simplex virus (HSV):

  1. Have history of oral or genital herpes and unable and/or unwilling to utilize prophylactic antiviral medication.
  2. Have a history of ocular herpes.
  3. Have active oral or genital herpes or are currently receiving treatment for HSV infection.
* Have complicating systemic diseases (e.g., medical conditions causing immunosuppression, active systemic infection) that would preclude the gene transfer or ocular surgery.
* Have known sensitivity or allergy to systemic corticosteroids or other immunosuppressive medications.
* Have used anti-coagulant agents that may alter coagulation
* Have received any vaccination/immunization within 28 days prior to screening and/or during screening with the exception of the influenza vaccine, which is only exclusionary if they have received the influenza vaccine within 28 days prior to randomization.
* Have used systemic corticosteroids or other immunosuppressive medications within 3 months prior to screening and/or intend to use during screening.
* Have previously received any AAV gene therapy product, stem cell therapy, cell-based therapy, or similar biologics.

Ocular Exclusion Criteria (Either Eye):

* Have pre-existing eye conditions that would preclude the planned surgery, interfere with the interpretation of study endpoints, or increase the risk of surgical complications
* Have significant media opacity impacting evaluation of the retina or vitreous.
* Had intraocular surgery within 90 days of study treatment administration.
* Have any active ocular/intraocular infection or inflammation
* Have a history of steroid-induced raised IOP of >25 mmHg following corticosteroid exposure, despite topical IOP-lowering pharmacologic therapy.
* Have any artificial retinal implant or prosthesis.
* Have absence of clear ocular media and/or inadequate pupil dilation to facilitate good quality OCT images.
* Have any history of rhegmatogenous retinal detachment.
* Have myopia (spherical equivalent) exceeding -10 diopters (or axial length of >30 mm if PI deems it appropriate to measure) or presence of pathologic myopia in the study eye.
* Have passed the Low Contrast Ora-VNC™ mobility course in either eye or binocularly at any screening visit.

Ages: 8 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of responding eyes between treated and control eyes in the low dose group and high dose group at 12 months, as measured by MAIA microperimetry, where response is defined as a 7dB or more improvement in at least 5 loci. | Day 0 - Month 12

SECONDARY OUTCOMES:
Proportion of responding eyes in treated eyes versus control eyes in the low dose group and the high dose group at Month 12 where responder is defined as an ORA-VNC mobility test score improvement of 2 or more luminance levels. | Day 0 - Month 12
Proportion of responding eyes in treated versus control eyes in the low dose group and the high dose group at Month 12, as measured by MAIA microperimetry, where responder is defined as a 7 dB or more improvement in at least 5 loci within bleb. | Day 0 - Month 12
Proportion of responding eyes in treated vs control eyes in the low dose group and the high dose group at Month 12, measured by MAIA microperimetry where responder is defined as 7 dB or more improvement in at least 5 loci within the central 16 loci | Day 0 - Month 12
Difference in mean change from baseline in the central 36 loci (C36) mean sensitivity, as measured by MAIA microperimetry, in treated eyes versus control eyes in the low dose group and high dose group at Month 12. | Day 0 - Month 12
Difference in mean change from baseline in "within bleb" mean sensitivity, as measured by MAIA microperimetry, in treated eyes versus control eyes in the low dose group and high dose group at Month 12. | Day 0 - Month 12
Difference in mean change from baseline in central 10 degrees of vision on light adapted static perimetry, as measured by Octopus 900, in treated eyes versus control eyes in the low dose group and high dose group at Month 12. | Day 0 - Month 12
Difference in mean change from baseline in BCVA, as measured by ETDRS or tumbling "E" chart, in treated eyes versus control eyes in the low dose group and high dose group at Month 12. | Day 0 - Month 12
Proportion of responding eyes in treated versus control eyes in the low dose group and high dose group at Month 12 where responder is defined as a 10-letter vision gain as measured by ETDRS or tumbling "E" chart. | Day 0 - Month 12
Difference in mean change from baseline in the EZ area, as measured by SD-OCT, in treated eyes versus control eyes in the low dose group and high dose group at Month 12 Visit. | Day 0 - Month 12
Mean change from baseline in Impact of Vision Impairment (IVI) (Weih et al, 2002; Lamoureaux et al, 2007) or Impact of Vision Impairment for Children (IVI-C) (Cochrane et al, 2008) in the low dose group and high dose group at Month 12 Visit | Day 0 - Month 12
Mean change from baseline in Patient Global Impressions of Change (PGI-C) and Patient Global Impressions of Severity (PGIS) in the low dose group and high dose group at Month 12 Visit. | Day 0 - Month 12

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Florida, Jacksonville, Florida
  - Boston Children's Hosptial, Boston, Massachusetts
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

REFERENCES:
- [Derived] Wang CY, Chen L, Lin TY, Huang SP. Systematic Identification of Candidate Genes for Inherited Retinal Disease Gene Therapy Integrating Worldwide IRD Cohort and Single-Cell Analysis. J Ophthalmol. 2025 Jun 12;2025:7014745. doi: 10.1155/joph/7014745. eCollection 2025. PMID 40547876